CLINICAL TRIAL: NCT01447693
Title: Treatment of Uremic Pruritus by Olive-omega 3 Ointment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130/06
Record Dates: First submitted 2007-12-31; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Uremic Pruritus
Keywords: uremia; pruritus; oliva-omega 3
MeSH Terms: conditions — Uremia; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: application of ointment (olive-omega 3 ointment)

SUMMARY:
Background.

Uremic pruritus is still a common phenomenon in patients with end-stage renal failure. It is regarded as one of the most bothersome symptoms in patients on chronic dialysis.

The pathogenesis of uremic itch remains unclear. Several theories have been proposed like dryness of the skin, imbalance in divalent ions, peripheral neuropathy and others.

Many treatment modalities have been tried to reduce uremic pruritus, however , the majority of them produced only temporary improvement. Therefore , every new therapeutic option for uremic pruritus is desirable.

This study will undertaken to evaluate the efficacy of a cream which included olive oil and omega-3 fatty acids.

Olive Omega-3 is an efficient product that soothes itchiness of cracked and very dry skin.

The product is unique and based on patented technology developed by the Technion Research and Development Foundation in Haifa.

Olive Omega-3 is an ointment composed of all natural ingredients. The main active ingredients are extra virgin olive oil , fish oil and vitamin C. The oils provides the skin with fatty acids that are vital for its proper functioning and help in the skin recovery. Sugar cane extract improves the skin's flexibility by removing dead cells and enhancing water retention in the upper layer of the skin.

When applied on clean skin , the product is quickly absorbed , producing a sensation of relief within a short time period. Treatment can be repeated as often as required with no limitations and its use is not contraindicative of any other medical treatment.

Patients and Methods.

About 20 patients on chronic hemodialysis suffering from uremic pruritus will be include in the study.

All patients will undergo dermatologic examination. All patients will be score by intensity of itching according to 3-point scale , as follows:

1. - patches of fine , powdery scales
2. - moderate scaling with beginning cracks
3. - intense scaling , moderate cracks The patients all applied Olive Omega-3 ointment for 50% of body and Vaseline ointment for the second one. The treatment will repeated twice daily for two weeks.

At the end of 2 weeks application global tolerance will evaluate using the following 3-point scale:

1. very good
2. good
3. poor

At the same time global agreement of the patients will evaluate according to the following scale :

1. - very satisfactory
2. - satisfactory 3- poorly satisfactory.

Statistical analysis will be performed by use of Wilcoxon test .

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients which have treated at least 3 months

Exclusion Criteria:

* Dermatologic diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)